CLINICAL TRIAL: NCT01882972
Title: Safety and Efficacy of Home-based Resistance Training in Colorectal Cancer Survivors
Brief Title: Strength for Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator left Loyola
Sponsor: Loyola University (Other)
Collaborators: Hygenic Corporation (Unknown)
Responsible Party: Principal Investigator, Kate Wolin, Associate Professor, Loyola University Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 205243
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Exercise; Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Exercise 12 week home-based resistance exercise training intervention. Participants will be coached to engage in resistance training 3 days per week and aerobic exercise for 30 minutes at least 5 days per week for 12 weeks.
  Interventions: Behavioral: Exercise
- control (Placebo Comparator): Participants in the attention control arm will not be asked to cease activity they already participate in but will be instructed not to begin a new exercise program for 12 weeks. Participants will receive a meditation CD to use daily to account for the time intervention arm participants are engaged in exercise.
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Exercise
  Other Names: Home-based exercise using Therabands
  Arms: Exercise
Behavioral: Meditation
  Other Names: A healing meditation for cancer patients CD
  Arms: control

SUMMARY:
Despite a robust literature on the benefits of exercise for cancer survivors, most of the research to date falls in two primary areas - aerobic exercise and breast cancer survivors. The focus on aerobic training alone is a concern as resistance training is critical for building the muscle mass necessary to maintain physical function. However, concerns have been raised about the potential for higher than tolerated adverse event rates during resistance training, particularly that which is unsupervised, despite a history of safe use of resistance training in other chronically diseased patient populations. The aim of this pilot study is to demonstrate the feasibility, safety and quality of life benefit of a home-based resistance-training program among colorectal cancer survivors. The investigators will recruit n=30 men and women with stage I-III colon cancer. Participants will be randomized to a home-based exercise intervention that combines aerobic and resistance exercise. Control arm participants will receive a home-based meditation program.

DETAILED DESCRIPTION:
The investigators will recruit n=30 patients with stage I-III colorectal cancer and randomize them to a 12-week resistance training intervention with Theraband and existing evidence- based materials or attention control using a meditation intervention. Using an electronic survey tool, patients will complete a baseline questionnaire on key outcomes (quality of life, fatigue, side effects) and potential confounders and will consent to a medical record review. These will also be assessed via at 4 weeks post randomization and 12 weeks post randomization. Participants in the intervention group will receive one-time in person instruction in the exercises derived from the existing evidence base of home-based resistance training programs for older adults and cancer survivors. They will be sent home with a book demonstrating the exercises, a log and a set of appropriate resistance bands. Weekly follow-up calls will occur for the duration of the intervention and updates on the call results will be provided to the colon cancer clinic nurse so that care is integrated. Participants in the attention control group will be mailed a meditation CD. Follow-up in the control group will parallel that of the intervention group, with weekly calls.

ELIGIBILITY:
Inclusion Criteria:

* stage I-III colorectal cancer
* completed surgical treatment
* at least 12 weeks post-surgery.
* at least 4 weeks post adjuvant therapy.
* age 18 and older.

Exclusion Criteria:

* patients who had surgery more than 24 months ago.
* patients with related pre-existing conditions (i.e., Crohn's disease, ulcerative colitis, familial polyposis syndromes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | 14 months
  Ability to meet the recruitment goal of 30 subjects in a 14 month period, reflecting a participation rate of at least 20% among approached and eligible patients
Retention feasibility | 14 months
  Retention of at least 80% of randomized patients to the follow-up visit. A drop-out rate of less than 20%

SECONDARY OUTCOMES:
Pain | 12 weeks
  Change in participant reported pain from baseline to 12 weeks
quality of life | 12 weeks
  Change in Quality of life score as measured by the FACT-C and FACT-F from baseline to 12 weeks
Surgical Complications | 12 weeks
  Difference in rate of reported surgical complications between arms at 12 weeks
Self-reported Exercise-related Injury | 12 weeks
  difference in self reported exercise-related injury rate between arms at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Wolin, ScD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Chicago, Maywood, Illinois, United States